CLINICAL TRIAL: NCT07017582
Title: Bicarbonate and Rugby
Brief Title: The Effect of Bicarbonate Supplementation on Performance and Gastrointestinal Symptoms in Rugby Players.
Acronym: Bicarbrugby
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Burgos (Other)
Collaborators: Universidad Isabel I (Unknown)
Responsible Party: Principal Investigator, MARIA MARTINEZ, Doctor, Universidad de Burgos
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Bicarbonaterugby; Bicarbonaterugby (Registry Identifier: Bicarbonaterugby)
Record Dates: First submitted 2025-05-23; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Supplementation
Keywords: Bicarbonate; Rugby; Performance

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bicarbonate (Active Comparator): Supplementation with 0.3 g/kg of sodium bicarbonate
  Interventions: Dietary Supplement: Soidum Bicarbonate
- Placebo (Placebo Comparator): Supplementation with placebo: 0.03 g·kg-1 body mass sodium chloride
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Soidum Bicarbonate — Supplementation with 0.03 g/kg of sodium bicarbonate
  Arms: Bicarbonate
Dietary Supplement: Placebo — 0.03 g·kg-1 body mass sodium chloride
  Arms: Placebo

SUMMARY:
The objetive of the study was to determine whether sodium bicarbonate supplementation improves athletic performance and/or reduces fatigue in elite rugby players.

The participants were 17 elite rugby players. Half of the participants receive sodium bicarbonate (0.3 g/kg body weight), the other half receive a placebo (salt). Ingestion of the supplementation/placebo occured 90 minutes before high-intensity rugby-specific training Variables analysed were measure at baseline, prior to exercise, during exercise and after exercise.

ELIGIBILITY:
Inclusion Criteria:

* Male rugby players who were competing in the First Spanish National League (Division de Honor A) voluntarily agreed to participate in the study after attending an informative session

Exclusion Criteria:

* injury or illness on test day

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-02-14 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Capillary blood lactate | At baseline (prior to supplementation), prior to exercise (immediately before beginning exercise protocol), after exercise (immediately after finishing exercise protocol).
  Lactate concentrations were measured in a capillary blood sample obtained fromparticipants' fingertips using a portable analyzer (Lactate 2, Arkray, Kyoto, Japan)

SECONDARY OUTCOMES:
Countermovement jump | At baseline (prior to supplementation) and after exercise (immediately after finishing exercise protocol).
  For the CMJ, subjects started from an upright position withhands on waist and then executed a countermovement jump by flexing the knees to 90◦and jumping as high as possible. During the flight stage, they were instructed to keep theirknees extended to 180◦, without hyperextending the hips . Jump height was measuredon an infrared platform (Optojump, Microgate, Bolzano, Italy).
Gastrointestinal (GI) symptoms | At baseline (before supplementation), prior to exercise (immediately before beginning exercise protocol), after exercise (immediately after finishing exercise protocol).
  Questionnaires consisted of nine 100-mm visual analog scales (VASs). The VASs were anchored at each end with no symptom on the left-hand side and severe symptom on the right-hand side. Participants were asked to rate the severity of their symptoms. If they were experiencing no symptoms, they circled the appropriate words, for example, no nausea. If they were experiencing some symptoms, they indicated their overall rating by placing a vertical mark on the line.
  The VASs were used to measure symptoms of nausea, flatulence, stomach cramping, belching, stomachache, bowel urgency, diarrhea, vomiting, and stomach bloating.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Burgos, Burgos, Spain

IPD SHARING:
Plan to Share IPD: No
Confidential data regarding a rugby club